CLINICAL TRIAL: NCT02640131
Title: A Bio-psychosocial Sexual Health Intervention for Prostate Cancer Survivors and Partners: a Feasibility Study
Acronym: BSHR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 701840; 701840 (Other Grant/Funding Number: Canadian Cancer Society Research Institute)
Record Dates: First submitted 2014-05-28; First posted 2015-12-28 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Prostate Cancer; Erectile Dysfunction; Sexual Dysfunction
Keywords: prostate cancer; radical prostatectomy; survivorship; quality of life; erectile dysfunction; sexual dysfunction; feasibility study
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BSHR Intervention (Experimental): Couples will attend 30-minute clinic consultations with an Urologist and a Sexual Health Counsellor and receive session-specific chapters of the Kindness, Intimacy, Sexuality and Satisfaction manual over the course of the intervention.
  The BSHR Intervention involves two complementary components; the bio-medical, and the psychosocial. The bio-medical component for both arms intervention includes an urologist consultation at a pre-operative appointment and 5 f/u appointments. Patients/partners are provided instruction on the use of pro-erectile agents/devices.
  The psychosocial component aims to support maintenance of intimacy, pro-erectile therapy use, and regular satisfying sexual activity. At each time point, participants receive sexual health counseling and manualized support.
  Interventions: Behavioral: Biomedical Component; Behavioral: Psychosocial Component
- Attention Control (Active Comparator): Survivorship Counseling: Couples will attend 30-minute clinic consultations with an Urologist and a Survivorship Counsellor (SurvC) and receive a Kegel Exercise booklet and receive appointment-specific chapters of the Challenging Prostate Cancer: "Nutrition, Exercise, and You Manual". The bio-medical component is the same in both arms.
  The core topics discussed during over 7 counseling sessions include: preparation for immediate post-surgery recovery, Kegel exercises, nutrition and prostate cancer, exercise and prostate cancer, and maintaining healthy lifestyle change.
  Interventions: Behavioral: Biomedical Component; Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Biomedical Component — Bio-medical: The bio-medical component includes an appointment with urologist pre-operatively and 5 follow-up appointments. Patients/partners are provided instruction on the use of pro-erectile agents/devices.
Behavioral: Psychosocial Component — Psychosocial: aims to support maintenance of intimacy, pro-erectile therapy use, and regular satisfying sexual activity. At each time point, participants receive standardized sexual health counselor (SexHC) counseling and manualized support.
  Arms: BSHR Intervention
Behavioral: Attention Control — Couples will attend 30-minute clinic consultations with an Urologist and a Survivorship Counsellor (SurvC) at 3-4, 7-8, and 12-13 months post radical prostatectomy (RP). Couples will receive a Kegel Exercise booklet and receive appointment-specific chapters of the Challenging Prostate Cancer: Nutrition, Exercise, and You (CPC) manual (a patient self-help manual written by the Princess Margaret Prostate Centre team). The core topics discussed during the counselling sessions include: preparation for immediate post-RP recovery, Kegel exercises, nutrition and prostate cancer (PC), exercise and PC, and maintaining healthy lifestyle change.
  Arms: Attention Control

SUMMARY:
The burden of sexual dysfunction after prostate cancer surgery is responsible for the single greatest impact on patient/partner health-related quality of life; substantially more so than concern for cancer recurrence, or any other post-surgery side-effect. Consequently, there is a great need for progressive and distributable sexual health rehabilitation interventions designed to uphold intimacy and optimal sexual health. If the biomedical-psychosocial intervention is ultimately found beneficial, it will result in: 1) an empirically-based intervention that helps patients/partners maintain optimal health-related quality of life after prostate cancer surgery, and 2) a highly structured protocol and manualized intervention that is translatable to other treatment groups (e.g. radiation therapy) and University/Community-based hospitals.

DETAILED DESCRIPTION:
Previous Research: The prevalence of sexual dysfunction (SD) after prostate cancer surgery, coupled with the severity of impact and lack of successful intervention, make SD one of the most substantial health-related quality of life burdens in all of cancer survivorship. In 2012, 21,000 men will be added to the pool of Canadian prostate cancer (PC) survivors. Approximately 70% of men will suffer SD post-surgery and 60% will experience significant distress in response to SD. Similarly, partners may experience even greater distress than patients. Research examining the nature of the distress reveals that the significance of SD extends beyond the ability to have an erection, and includes guilt, depression, anxiety, anger, and reductions in intimacy. Unfortunately, there are no reported interventions that have been successful in reducing the impact of SD on long term couple health-related quality of life.

Project Description: Men and their partners need an effective intervention to help them adapt to sexual dysfunction following prostate cancer surgery. In addressing this need we propose an innovative biomedical-psychosocial Intervention that emphasizes: 1) multidisciplinary intervention teams; 2) the active participation of the partner; and 3) a broad-spectrum medical, psychological, and social approach. The treatment goal of the intervention is to promote intimacy and optimal sexual health in affected couples. This is a preliminary study designed to determine the feasibility of running a large scale randomized controlled trial comparing the new biomedical-psychosocial intervention to an attention control condition.

Impact and Relevance: The burden of sexual dysfunction after prostate cancer surgery is responsible for the single greatest impact on patient/partner health-related quality of life; substantially more so than concern for cancer recurrence, or any other post-surgery side-effect. Consequently, there is a great need for progressive and distributable sexual health rehabilitation interventions designed to uphold intimacy and optimal sexual health. If the biomedical-psychosocial intervention is ultimately found beneficial, it will result in: 1) an empirically-based intervention that helps patients/partners maintain optimal health-related quality of life after prostate cancer surgery, and 2) a highly structured protocol and manualized intervention that is translatable to other treatment groups (e.g. radiation therapy) and University/Community-based hospitals.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for a Radical Prostatectomy at the Princess Margaret Cancer Centre(open, laparoscopic, robotic) for the first-line treatment of prostate cancer regardless of clinical stage of disease
* are hormone and/or chemotherapy-naïve
* have a sexual partner (heterosexual or homosexual) for at least the past 6 months
* are 18 years of age or older
* Partners of men who meet the above criteria and are 18 years of age or older

Exclusion Criteria:

* the patient or partner lacks English proficiency
* the patient is on nitrate therapy or has other contra-indications to phosphodiesterase type 5 inhibitors (PDE5i's)
* the patient does not have a sexual partner
* the patient or partner has a medical condition that would preclude safe sexual activity
* the patient has had previous treatment for PC
* the patient has previously and regularly used sexual aids/devices during the course of sexual activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-01; Primary Completion 2017-01 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Miller Social Intimacy Scale (MSIS) | At least 1 week prior to radical prostatectomy; 13-14 months post-radical prostatectomy
  Miller Social Intimacy Scale (MSIS):MSIS is a 17-item measure of the maximum level of intimacy currently experienced is used in this study. Each question has a scale of 1-10 with a higher score representing higher level of intimacy.

SECONDARY OUTCOMES:
International Index of Erectile Function (IIEF) | At least one week prior to radical prostatectomy; 13-14 months post-radical prostatectomy
  International Index of Erectile Function (IIEF) is validated as a brief, easily administered, patient-reported diagnostic tool for men as a measure for male optimal sexual health for Bio-medical Responders and Bio-medical Non-Responders. IIEF has 15 items in all with a scale from 0(1) to 5. Higher number indicates a better sexual function.
Female Sexual Function Inventory (FSFI) | At least one week prior to radical prostatectomy; 13-14 months post-radical prostatectomy
  Female Sexual Function Inventory (FSFI): the FSFI is a brief, 19-item self-report measure of female sexual function that provides scores on six domains of sexual function (Desire, Arousal, Lubrication, Orgasm, Satisfaction, Pain) as well as a total score. The full scale score is obtained by adding the six domain scores. It should be noted that within the individual domains, a domain score of zero indicates that no sexual activity was reported during the past month. Higher score indicates a better sexual function.
Hospital Anxiety and Depression Scale (HADS) | At least one week prior to radical prostatectomy; 13-14 months post-radical prostatectomy
  Hospital Anxiety and Depression Scale (HADS) is used to determine the levels of anxiety and depression that participants are experiencing. The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each question has a scale of 0 to 3 and the total score can be calculated for the two domains (anxiety and depression) by adding the scores together. For each domain, a score of 0-7 = Normal level of anxiety/depression; a score of 8-10 = borderline case of anxiety/depression; 11-21 = case of anxiety/depression.
Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) | 13-14 months post-radical prostatectomy
  Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) is used to measure participants' satisfaction with Erectile Dysfunction Treatment. EDITS has 11 items with a scale from 1 to 5. Higher number indicates a higher satisfaction level.
Sexual Health Rehabilitation Record | 3-4 months post-radical prostatectomy;7-8 months post-radical prostatectomy;12-13 months post-radical prostatectomy
  *investigator designed
Expanded Prostate Cancer Index Composite (EPIC) | At least 1 week prior to radical prostatectomy; 13-14 months post-radical prostatectomy
  EPIC is a comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment. The version we used contains 26 item and the 5 domains: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal. Response options for each EPIC item form a Likert scale, and multi-itemscale scores are transformed linearly to a 0-100 scale, with higher scores representing better HRQOL (Health-Related Quality of Life).designed to evaluate patient function and bother after prostate cancer treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Matthew, PhD, C.Psych, Principal Investigator — University Health Network, Toronto
Locations (1):
- The Prostate Centre, Princess Margaret Hospital, Toronto, Ontario, Canada